CLINICAL TRIAL: NCT07228039
Title: A Double-Blind Prospective RCT Assessment of ESP Blocks for Analgesia Following Posterior Spinal Fusion
Brief Title: ESP Blocks for Posterior Spinal Fusion
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00118950
Record Dates: First submitted 2025-11-12; First posted 2025-11-13 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Postoperative Pain
Keywords: ESP Block; Spinal Fusion; Multimodal Analgesia
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- ESP + Liposomal Bupivacaine (Experimental): Group 1 receives ESP block with 0.5% bupivacaine plus liposomal bupivacaine.
  Interventions: Drug: ESP Block with Bupivacaine + Liposomal Bupivacaine
- ESP + Plain Bupivacaine (Experimental): Group 2 receives ESP block with 0.5% plain bupivacaine.
  Interventions: Drug: ESP Block with Bupivacaine

INTERVENTIONS:
Drug: ESP Block with Bupivacaine — Cervical and lumbar ESP blocks performed under ultrasound guidance using plain bupivacaine.
  Arms: ESP + Plain Bupivacaine
Drug: ESP Block with Bupivacaine + Liposomal Bupivacaine — Cervical and lumbar ESP blocks performed under ultrasound guidance using bupivacaine admixed with liposomal bupivacaine.
  Arms: ESP + Liposomal Bupivacaine

SUMMARY:
This prospective randomized double-blind study evaluates the efficacy of erector spinae plane (ESP) blocks on postoperative pain in patients undergoing cervical or lumbar posterior spinal fusion. Patients will receive either 0.5% bupivacaine plus liposomal bupivacaine or 0.5% plain bupivacaine. Outcomes include opioid consumption over 72 hours, pain scores, length of stay, and time to ambulation.

ELIGIBILITY:
Inclusion Criteria

* English speaking
* Age 18-75
* ASA physical status 1-3
* Undergoing elective cervical or lumbar posterior spinal fusion (≤3 levels)

Exclusion Criteria

* Age <18 or >75
* ASA IV or V
* Non-English speaking
* BMI >40
* Opioid dependence
* Chronic pain
* Anticoagulation or coagulopathy
* Injection site infection
* Hepatic or renal insufficiency
* Allergy to study drugs
* Pregnancy
* Inability to communicate with investigators

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain as measured by opiate consumption | 72 hours
  Morphine MilliEquivalents

SECONDARY OUTCOMES:
Postoperative Pain at rest and with movement as measured by patient reported pain scores | 4, 8, 12, 24, 48, and 72 hours
  Numeric Rating Scale (0-10)
Discharge Readiness | 72 hours
  Hospital and PACU Length of Stay
Postoperative Pain Severity as measured by required time for patient controlled-analgesia | 72 hours
  Duration of patient controlled analgesia use
Incidents of post-operative nausea and vomiting | 72 hours
  Post-operative Nausea and Vomiting
Time to first ambulation | 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Davies, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No